CLINICAL TRIAL: NCT04303078
Title: Quantifying Energetic Demands of Walking for People With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Gillette Children's Specialty Healthcare (Other)
Responsible Party: Principal Investigator, Katherine Steele, Associate Professor, Engineering, University of Washington
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00014591; R21HD104112 (NIH)
Record Dates: First submitted 2020-02-21; First posted 2020-03-10 (Actual); Results first posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Cerebral Palsy
Keywords: Energetic cost
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Children with Cerebral Palsy (Cases) (Experimental): Children meeting inclusion/exclusion criteria with a diagnosis of cerebral palsy.
  Interventions: Other: Varying levels of harness support during walking
- Typically Developing Children (Controls) (Other): Children meeting inclusion/exclusion criteria without a diagnosis of cerebral palsy or other condition.
  Interventions: Other: Varying levels of harness support during walking

INTERVENTIONS:
Other: Varying levels of harness support during walking — Participants will complete a standard gait and motion analysis at varying levels of harness support and stabilization (low, moderate, and high levels).

SUMMARY:
The purpose of this study is to examine the underlying mechanisms that contribute to high energy costs for people with cerebral palsy (CP) as they walk.

The investigators will characterize the cost landscape of children with CP, quantifying the magnitude of cost (net nondimensional oxygen consumption) associated with walking and common sub-tasks of walking, such as supporting and stabilizing the body.

DETAILED DESCRIPTION:
Children with CP use large amounts of energy to walk and move, leading to fatigue and limiting participation. For people with CP the energetic cost of walking is on average over two times higher than typically-developing (TD) peers. This means that for people with CP, walking is as tiring as jogging or climbing stairs. An energetic cost of this magnitude restricts activities of daily living (ADL) and causes exhaustion.

While the investigators and many others have sought to reduce these energetic costs through surgical interventions, rehabilitation, orthotics, or other assistive devices, these strategies have failed to result in meaningful reductions in energy. To design strategies that successfully reduce walking costs, the investigators must first understand the underlying mechanisms contributing to elevated cost in people with CP. This basic-science research will provide the foundation to create evidence-based strategies to decrease energy costs, minimize fatigue, and increase quality of life for people with CP and other neurologic injuries.

ELIGIBILITY:
Inclusion Criteria for Cases:

* 8-17 years old
* Diagnosed with bilateral cerebral palsy
* Gross Motor Function Classification System II
* No surgery within the last 9 months
* No current baclofen pump or explantation in the last 2 months
* No botulinum toxin or phenol injections in the last 2 months
* Had a prior gait and motion analysis at Gillette Children's Specialty Healthcare
* Participant and caregiver able to speak and read English
* Ability to follow instructions

Inclusion Criteria for Controls:

* 8-17 years old
* Participant and caregiver able to speak and read English
* Ability to follow instructions

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2023-08-15 (Actual); Primary Completion 2025-06-17 (Actual); Study Completion 2025-06-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Steele, PhD, Principal Investigator — University of Washington; Michael Schwartz, PhD, Principal Investigator — Gillette Children's Specialty Healthcare
Locations (1):
- Gillette Children's Specialty Healthcare, Saint Paul, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Campbell J, Ball J. Energetics of walking in cerebral palsy. Orthop Clin North Am. 1978 Apr;9(2):374-7. No abstract available. PMID 662304

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited through Gillette Children's via electronic medical record search, flyers, social media postings, and word of mouth at local clinics and community organizations. Recruitment started in the Summer of 2023, after a delay due to a facility flood, and was completed in the Summer of 2025.
Period: Overall Study
Arm/Group | Children With Cerebral Palsy (Cases) | Typically Developing Children (Controls)
Started | 24 | 10
Completed | 23 | 10
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: The sample size was based on differences in costs between cerebral palsy and typically-developing groups from retrospective analyses and literature. The statistical plan was designed to detect a similar difference in cost between groups with a 3:1 allocation with alpha = 0.05 and 90% power, with a required sample size of 21 children with CP and 7 typically-developing peers stratified by age and sex.
Groups:
- Total: Total of all reporting groups
Arm/Group | Children With Cerebral Palsy (Cases) | Typically Developing Children (Controls) | Total
Number analyzed (Participants) | 24 | 10 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.8 (3.0) | 12.8 (2.9) | 12.8 (2.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 5 | 14
  Male | 15 | 5 | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 22 | 10 | 32
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 23 | 9 | 32
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Net Nondimensional Oxygen Cost
Description: Steady-state net nondimensional oxygen consumption while walking on a treadmill. Percent change in oxygen consumption was evaluated between baseline without support and with vertical and lateral support.
Time Frame: Baseline walking trial with harness on (5-minutes) and support walking trials with vertical or lateral support in harness system (5-minutes)
Population: One participant with cerebral palsy consented, but did not participate in the protocol. Issues with the system precluded inclusion of 9 additional participants with cerebral palsy for the lateral support analysis.
Measure: Mean (Standard Deviation); unit: Percent change relative to baseline
Arm/Group | Children With Cerebral Palsy (Cases) | Typically Developing Children (Controls)
Number analyzed (Participants) | 23 | 10
Percent change relative to baseline
  Percent Change (Vertical Support) | -34.13 (21.45) | -15.86 (17.76)
  Percent Change (Lateral Support): number analyzed (Participants) | 14 | 10
  Percent Change (Lateral Support) | 1.07 (7.07) | -0.60 (10.19)

2. Secondary Outcome: Three-dimensional Gait Kinematics (Baseline)
Description: Five features describing kinematics during gait in the harness system without vertical or lateral support collected from marker-based motion capture. Since the harness system differed between vertical and lateral support, baseline kinematics are reported separately for each system in the rows below. The features include (1) median pelvic tilt during the stance phase, (2) peak hip extension, (3) peak knee extension, (4) peak ankle plantarflexion, and (5) the foot progression angle relative to fore-aft direction.
Time Frame: Initial trial without support (5-minutes)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Children With Cerebral Palsy (Cases) | Typically Developing Children (Controls)
Number analyzed (Participants) | 23 | 10
Degrees
  Median Stance Pelvic Tilt (Vertical Support - Baseline) | 21.6 (8.0) | 13.6 (6.6)
  Median Stance Pelvic Tilt (Lateral Support - Baseline): number analyzed (Participants) | 14 | 10
  Median Stance Pelvic Tilt (Lateral Support - Baseline) | 23.4 (9.2) | 16.2 (7.6)
  Peak Stance Hip Extension (Vertical Support - Baseline) | 24.3 (11.5) | 13.2 (7.4)
  Peak Stance Hip Extension (Lateral Support - Baseline): number analyzed (Participants) | 14 | 10
  Peak Stance Hip Extension (Lateral Support - Baseline) | 27.1 (12.0) | 16.5 (9.5)
  Peak Stance Knee Extension (Vertical Support - Baseline) | 14.1 (12.9) | 0.1 (3.8)
  Peak Stance Knee Extension (Lateral Support - Baseline): number analyzed (Participants) | 14 | 10
  Peak Stance Knee Extension (Lateral Support - Baseline) | 13.3 (10.2) | 0.5 (6.8)
  Peak Stance Ankle Plantarflexion (Vertical Support - Baseline) | -1.2 (8.7) | -6.1 (2.4)
  Peak Stance Ankle Plantarflexion (Lateral Support - Baseline): number analyzed (Participants) | 14 | 10
  Peak Stance Ankle Plantarflexion (Lateral Support - Baseline) | -0.8 (6.9) | -5.3 (3.4)
  Median Stance Foot Progression (Vertical Support - Baseline) | -5.7 (10.1) | -5.6 (10.2)
  Median Stance Foot Progression (Lateral Support - Baseline): number analyzed (Participants) | 14 | 10
  Median Stance Foot Progression (Lateral Support - Baseline) | -6.2 (9.0) | -5.4 (10.5)

3. Secondary Outcome: Three-dimensional Gait Kinematics (Support)
Description: Five features describing kinematics during gait in the harness system with vertical and lateral support. The features include (1) median pelvic tilt during the stance phase, (2) peak hip extension, (3) peak knee extension, (4) peak ankle plantarflexion, and (5) the foot progression angle relative to fore-aft direction.
Time Frame: Trial with maximum support (5-minutes)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Children With Cerebral Palsy (Cases) | Typically Developing Children (Controls)
Number analyzed (Participants) | 23 | 10
Degrees
  Median Stance Pelvic Tilt (Maximum Vertical Support) | 22.1 (9.5) | 18.0 (6.7)
  Median Stance Pelvic Tilt (Maximum Lateral Support): number analyzed (Participants) | 14 | 10
  Median Stance Pelvic Tilt (Maximum Lateral Support) | 23.0 (8.3) | 16.4 (8.3)
  Peak Stance Hip Extension (Maximum Vertical Support) | 21.5 (11.9) | 15.4 (8.3)
  Peak Stance Hip Extension (Maximum Lateral Support): number analyzed (Participants) | 14 | 10
  Peak Stance Hip Extension (Maximum Lateral Support) | 28.0 (10.1) | 16.1 (9.9)
  Peak Stance Knee Extension (Maximum Vertical Support) | 13.0 (12.9) | 1.8 (7.8)
  Peak Stance Knee Extension (Maximum Lateral Support): number analyzed (Participants) | 14 | 10
  Peak Stance Knee Extension (Maximum Lateral Support) | 15.0 (8.8) | 0.4 (5.3)
  Peak Stance Ankle Plantarflexion (Maximum Vertical Support) | -2.0 (9.4) | -4.9 (5.2)
  Peak Stance Ankle Plantarflexion (Maximum Lateral Support): number analyzed (Participants) | 14 | 10
  Peak Stance Ankle Plantarflexion (Maximum Lateral Support) | -0.1 (6.9) | -5.1 (2.1)
  Median Stance Foot Progression (Maximum Vertical Support) | -4.1 (10.9) | -3.9 (8.9)
  Median Stance Foot Progression (Maximum Lateral Support): number analyzed (Participants) | 14 | 10
  Median Stance Foot Progression (Maximum Lateral Support) | -6.5 (9.7) | -8.5 (8.2)

4. Secondary Outcome: Three-dimensional Gait Kinetics (Baseline)
Description: Three features describing kinetics during gait in the harness system without vertical or lateral support collected from marker-based motion capture and instrumented treadmill for ground reaction forces. Since the harness system differed between vertical and lateral support, baseline kinematics are reported separately for each system in the rows below. The features include (1) peak hip extensor moment, (2) peak knee extensor moment, and (3) peak ankle plantarflexor moment.
Time Frame: Initial trial without support (5-minutes)
Population: One participant with cerebral palsy consented, but did not participate in the protocol. Issues with the system precluded inclusion of 9 additional participants with cerebral palsy for the lateral support analysis. For kinetics, adequate force pate data was not acquired for one additional child with cerebral palsy during vertical support, as well as two children with cerebral palsy and three typically-developing children during lateral support.
Measure: Mean (Standard Deviation); unit: Nm/kg
Arm/Group | Children With Cerebral Palsy (Cases) | Typically Developing Children (Controls)
Number analyzed (Participants) | 23 | 10
Nm/kg
  Peak Hip Extensor Moment (Vertical Support - Baseline): number analyzed (Participants) | 22 | 10
  Peak Hip Extensor Moment (Vertical Support - Baseline) | 0.462 (0.156) | 0.604 (0.153)
  Peak Hip Extensor Moment (Lateral Support - Baseline): number analyzed (Participants) | 12 | 7
  Peak Hip Extensor Moment (Lateral Support - Baseline) | 0.447 (0.122) | 0.613 (0.255)
  Peak Knee Extensor Moment (Vertical Support - Baseline): number analyzed (Participants) | 22 | 10
  Peak Knee Extensor Moment (Vertical Support - Baseline) | 0.160 (0.132) | 0.321 (0.095)
  Peak Knee Extensor Moment (Lateral Support - Baseline): number analyzed (Participants) | 12 | 7
  Peak Knee Extensor Moment (Lateral Support - Baseline) | 0.119 (0.097) | 0.306 (0.158)
  Peak Ankle Plantarflexor Moment (Vertical Support - Baseline): number analyzed (Participants) | 22 | 10
  Peak Ankle Plantarflexor Moment (Vertical Support - Baseline) | 0.026 (0.032) | 0.068 (0.035)
  Peak Ankle Plantarflexor Moment (Lateral Support - Baseline): number analyzed (Participants) | 12 | 7
  Peak Ankle Plantarflexor Moment (Lateral Support - Baseline) | 0.033 (0.028) | 0.074 (0.038)

5. Secondary Outcome: Three-dimensional Gait Kinetics (Support)
Description: Three features describing kinetics during gait in the harness system with vertical and lateral support. . Since the harness system differed between vertical and lateral support, baseline kinematics are reported separately for each system in the rows below. The features include (1) peak hip extensor moment, (2) peak knee extensor moment, and (3) peak ankle plantarflexor moment.
Time Frame: Trial with maximum support (5-minutes)
Population: One participant with cerebral palsy consented, but did not participate in the protocol. Issues with the system precluded inclusion of 9 additional participants with cerebral palsy for the lateral support analysis. For kinetics, adequate force pate data was not acquired for two children with cerebral palsy during vertical support, as well as one typically-developing child during lateral support.
Measure: Mean (Standard Deviation); unit: Nm/kg
Arm/Group | Children With Cerebral Palsy (Cases) | Typically Developing Children (Controls)
Number analyzed (Participants) | 23 | 10
Nm/kg
  Peak Hip Extensor Moment (Maximum Vertical Support): number analyzed (Participants) | 21 | 10
  Peak Hip Extensor Moment (Maximum Vertical Support) | 0.269 (0.046) | 0.312 (0.104)
  Peak Hip Extensor Moment (Maximum Lateral Support): number analyzed (Participants) | 14 | 9
  Peak Hip Extensor Moment (Maximum Lateral Support) | 0.465 (0.119) | 0.559 (0.152)
  Peak Knee Extensor Moment (Maximum Vertical Support): number analyzed (Participants) | 21 | 10
  Peak Knee Extensor Moment (Maximum Vertical Support) | 0.103 (0.052) | 0.177 (0.053)
  Peak Knee Extensor Moment (Maximum Lateral Support): number analyzed (Participants) | 14 | 9
  Peak Knee Extensor Moment (Maximum Lateral Support) | 0.122 (0.133) | 0.302 (0.092)
  Peak Ankle Plantarflexor Moment (Maximum Vertical Support): number analyzed (Participants) | 21 | 10
  Peak Ankle Plantarflexor Moment (Maximum Vertical Support) | 0.012 (0.016) | 0.035 (0.027)
  Peak Ankle Plantarflexor Moment (Maximum Lateral Support): number analyzed (Participants) | 14 | 9
  Peak Ankle Plantarflexor Moment (Maximum Lateral Support) | 0.026 (0.031) | 0.056 (0.031)

6. Secondary Outcome: Passive Joint Range of Motion
Description: Compare passive joint range of motion (degrees) measured by lower extremity physical exam
Time Frame: One-time research visit (15 minutes)
Population: One participant with cerebral palsy consented, but did not participate in the protocol.
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Children With Cerebral Palsy (Cases) | Typically Developing Children (Controls)
Number analyzed (Participants) | 23 | 10
Degrees
  Popliteal Angle | 51.478 (11.747) | 34.000 (9.416)
  Maximum Knee Extension | -0.435 (6.940) | -4.700 (4.523)
  Knee Extensor Lag | 3.174 (6.336) | 0.000 (0.000)
  Maximum Ankle Dorsiflexion | 4.043 (6.725) | 13.200 (4.341)

7. Secondary Outcome: Selective Motor Control
Description: Selective motor control (0 patterned movement - 2 complete isolated movement)
Time Frame: One-time research visit (15 minutes)
Population: One participant with cerebral palsy consented, but did not participate in the protocol.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Children With Cerebral Palsy (Cases) | Typically Developing Children (Controls)
Number analyzed (Participants) | 23 | 10
Units on a Scale
  Hip Flexion | 1.348 (0.487) | 2.000 (0.000)
  Hip Extension | 1.826 (0.388) | 2.000 (0.000)
  Knee Extension | 1.870 (0.458) | 2.000 (0.000)
  Ankle Plantarflexion | 1.565 (0.662) | 2.000 (0.000)

8. Secondary Outcome: Lower Extremity Strength
Description: Lower extremity strength measures by the manual muscle test (0 no muscle contraction - 5 typical muscle function)
Time Frame: One-time research visit (15 minutes)
Population: One participant with cerebral palsy consented, but did not participate in the protocol.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Children With Cerebral Palsy (Cases) | Typically Developing Children (Controls)
Number analyzed (Participants) | 23 | 10
Units on a Scale
  Back Extensor Strength | 4.391 (1.076) | 5.000 (0.000)
  Hip Extensor Strength | 3.652 (1.071) | 5.000 (0.000)
  Knee Extensor Strength | 4.913 (0.417) | 5.000 (0.000)
  Plantarflexor Strength | 3.130 (1.325) | 5.000 (0.000)

ADVERSE EVENTS:
Time Frame: During a single visit, up to 3 hours.
Arm/Group | Children With Cerebral Palsy (Cases) | Typically Developing Children (Controls)
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/10
Other Adverse Events (participants affected / at risk) | 0/24 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-11-03): https://cdn.clinicaltrials.gov/large-docs/78/NCT04303078/Prot_SAP_000.pdf